CLINICAL TRIAL: NCT03922607
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ABBV-157 in Healthy Volunteers and in Subjects With Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Tolerability of ABBV-157 in Healthy Volunteers and in Participants With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M17-238
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Psoriasis
Keywords: Psoriasis; Chronic Plaque Psoriasis; ABBV-157; Healthy Volunteers
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Substudy 2: Group 2 (Experimental): Participants with chronic plaque psoriasis will be administered with ABBV-157 dose D or matching placebo on Day 1 through Day 28
  Interventions: Drug: ABBV-157; Drug: Placebo for ABBV-157
- Substudy 2: Group 1 (Experimental): Participants with chronic plaque psoriasis will be administered with ABBV-157 dose C or matching placebo on Day 1 through Day 28
  Interventions: Drug: ABBV-157; Drug: Placebo for ABBV-157
- Substudy 1: Group 3 (Experimental): Participants, who are healthy volunteers, will be administered with ABBV-157 dose C or matching placebo on Day 1 through Day 14
  Interventions: Drug: ABBV-157; Drug: Placebo for ABBV-157
- Substudy 1: Group 2 (Experimental): Participants, who are healthy volunteers, will be administered with ABBV-157 dose B or matching placebo on Day 1 through Day 14
  Interventions: Drug: ABBV-157; Drug: Placebo for ABBV-157
- Substudy 1: Group 1 (Experimental): Participants, who are healthy volunteers, will be administered with ABBV-157 dose A or matching placebo on Day 1 through Day 14
  Interventions: Drug: ABBV-157; Drug: Placebo for ABBV-157

INTERVENTIONS:
Drug: ABBV-157 — ABBV-157 will be administered orally as capsule
Drug: Placebo for ABBV-157 — Placebo for ABBV-157 will be administered orally as capsule

SUMMARY:
This is a study to evaluate pharmacokinetics (PK), safety and tolerability of ABBV-157 in healthy volunteers and in participants with chronic plaque psoriasis, and to evaluate the efficacy of ABBV-157 in the participants with psoriasis. This study consists of two substudies. Substudy 1 is a randomized, double-blind, placebo-controlled evaluation of multiple ascending oral doses of ABBV-157 in healthy adult volunteers. Substudy 2 is a randomized, double-blind, placebo-controlled study in which participants with moderate to severe chronic plaque psoriasis will be administered multiple oral doses of ABBV-157.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer should be between 18 and 55 years of age and in general good health for Substudy 1 and participant with moderate to severe chronic plaque psoriasis between 18 and 75 years of age for Substudy 2 at the time of enrollment.
* Participant should meet the laboratory assessments as mentioned in the protocol.

Exclusion Criteria:

* Participant has a history of epilepsy, any significant cardiac, respiratory, renal, hepatic, gastrointestinal, opthalmologic, hematologic,or psychiatric disease or disorder, or any uncontrolled medical illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Substudy 1: Cmax of ABBV-157 | Up to approximately 14 days
  Maximum observed plasma concentration (Cmax) of ABBV-157
Substudy 1: Tmax of ABBV-157 | Up to approximately 14 days
  Time to maximum observed plasma concentration (Tmax) of ABBV-157
Substudy 1: AUC0-24 Post-dose of ABBV-157 | Day 1
  Area under the plasma concentration-time curve from 0 to 24 hours (AUC0-24) post-dose of ABBV-157.
Substudy 1: Trough Concentration (Ctrough) of ABBV-157 | Up to approximately 14 days
  Observed Plasma Concentration at the End of the Dosing Interval (Ctrough) of ABBV-157
Substudy 1: AUCtau of ABBV-157 | Up to approximately 14 days
  The area under the plasma concentration-time curve over a dosing interval of tau (AUCtau).
Substudy 1: Apparent Oral Clearance (CL/F) | Day 14
  Clearance is defined as the volume of plasma cleared of the drug per unit time.
Substudy 1: Volume of Distribution (Vβ/F) | Day 14
  Volume of Distribution (Vβ/F) of ABBV-157
Substudy 1: Apparent Terminal Phase Elimination Constant (β) | Day 14
  Apparent Terminal phase elimination rate constant (β or Beta)
Substudy 1: Elimination Half-Life (t1/2) | Day 14
  Terminal phase elimination half-life (t1/2) of ABBV-157
Substudy 1: Fraction Excreted Unchanged in Urine (fe) | Day 14
  Fraction excreted unchanged in urine (fe)
Substudy 1: Apparent Renal Clearance (CLR) | Day 14
  Apparent Renal Clearance (CLR) of ABBV-157
Substudy 1: Accumulation ratio for Cmax | Up to approximately 14 days
  Accumulation ratio for Cmax
Substudy 1: Accumulation Ratio for AUCtau | Up to approximately 14 days
  Accumulation Ratio for AUCtau
Substudy 2: Cmax of ABBV-157 | Up to approximately 28 days
  Maximum observed plasma concentration (Cmax) of ABBV-157
Substudy 2: Tmax of ABBV-157 | Up to approximately 28 days
  Time to maximum observed plasma concentration (Tmax) of ABBV-157
Substudy 2: AUC0-24 Post-dose of ABBV-157 | Day 1
  Area under the plasma concentration-time curve from 0 to 24 hours (AUC0-24) post-dose of ABBV-157.
Substudy 2: AUCtau of ABBV-157 | Day 28
  The area under the plasma concentration-time curve over a dosing interval of tau (AUCtau)
Substudy 2: Apparent Oral Clearance (CL/F) | Day 28
  Clearance is defined as the volume of plasma cleared of the drug per unit time.
Substudy 2: Volume of Distribution (Vβ/F) | Day 28
  Volume of Distribution (Vβ/F) of ABBV-157
Substudy 2: Apparent Terminal Phase Elimination Constant (β) | Day 28
  Apparent Terminal phase elimination rate constant (β or Beta)
Substudy 2: Elimination Half-Life (t1/2) | Day 28
  Terminal phase elimination half-life (t1/2) of ABBV-157
Substudy 2: Accumulation ratio for Cmax | Up to approximately 28 days
  Accumulation ratio for Cmax
Substudy 2: Accumulation Ratio for AUCtau | Up to approximately 28 days
  Accumulation Ratio for AUCtau
Substudy 2: Trough Concentration (Ctrough) of ABBV-157 | Up to approximately 28 days
  Observed Plasma Concentration at the End of the Dosing Interval (Ctrough) of ABBV-157
Substudy 2: Percent Change in Psoriasis Area and Severity Index (PASI) score from Baseline | Up to approximately 28 days
  Psoriasis Area and Severity Index (PASI) score quantitative assessment of psoriasis disease state based on the amount of body surface area that is affected and the degree of severity.
Substudy 2: Change in Self-Assessment of Psoriasis Symptoms (SAPS) Score from Baseline | Up to approximately 28 days
  SAPS is a self-assessment questionnaire of psoriasis symptoms.
Number of Participants With Adverse Events (AEs) | Up to Day 58
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (10):
  - Total Skin and Beauty Derm Ctr /ID# 222593, Birmingham, Alabama
  - Alliance Dermatology and MOHs /ID# 222622, Phoenix, Arizona
  - Anaheim Clinical Trials LLC /ID# 213645, Anaheim, California
  - Dermatology Res. Assoc., CA /ID# 224980, Los Angeles, California
  - Providence Clinical Research /ID# 213339, North Hollywood, California
  - Advanced Medical Research /ID# 216090, Sandy Springs, Georgia
  - Acpru /Id# 213639, Grayslake, Illinois
  - University of Pittsburgh MC /ID# 224699, Pittsburgh, Pennsylvania
  - PPD PH I Clinical Unit /ID# 213062, Austin, Texas
  - Center for Clinical Studies - Webster TX /ID# 217352, Webster, Texas

IPD SHARING:
Plan to Share IPD: No